CLINICAL TRIAL: NCT00724048
Title: A Multi-center, North American, Randomized, Double-blind, Parallel Group Study Comparing Three Doses of ACR16 Versus Placebo for the Symptomatic Treatment of Huntington Disease (HART)
Brief Title: A Study of Pridopidine (ACR16) for the Treatment of Participants With Huntington's Disease
Acronym: HART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACR16 C009
Record Dates: First submitted 2008-07-24; First posted 2008-07-29 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-07

CONDITIONS: Huntington Disease
Keywords: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive a placebo capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), placebo capsule will be taken twice daily (BID) as 2 separate doses.
  Interventions: Other: Placebo
- ACR16 10 mg BID (Experimental): Participants will receive ACR16 10 milligrams (mg) capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 10 mg capsule will be taken twice daily (BID) as 2 separate doses (total dose: 20 mg).
  Interventions: Drug: ACR16
- ACR16 22.5 mg BID (Experimental): Participants will receive ACR16 22.5 mg capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 22.5 mg capsule will be taken twice daily (BID) as 2 separate doses (total dose: 45 mg).
  Interventions: Drug: ACR16
- ACR16 45 mg BID (Experimental): Participants will receive ACR16 45 mg capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 45 mg capsule will be taken twice daily (BID) as 2 separate doses (total dose: 90 mg).
  Interventions: Drug: ACR16

INTERVENTIONS:
Drug: ACR16 — ACR16 will be administered per dose and schedule specified in the arm description.
  Other Names: pridopidine
  Arms: ACR16 10 mg BID; ACR16 22.5 mg BID; ACR16 45 mg BID
Other: Placebo — Placebo matching to ACR16 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ACR16 is effective and safe in the symptomatic treatment of Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written Informed Consent prior to any study related procedure, including consent to genotyping of the CYP2D6 gene.
* Clinical features of HD, and a positive family history and/or the presence of ≥ 36 CAG repeats in the Huntington gene.
* Male or female age ≥ 30 years.
* Willing and able to take oral medication and to comply with the study specific procedures.
* Ambulatory, being able to travel to the assessment center, and judged by the Investigator as likely to be able to continue to travel for the duration of the study.
* Availability of a caregiver or family member to accompany the participant to two visits.
* A sum of ≥ 10 points on the mMS at the screening visit.
* For participants taking allowed antidepressants or other psychotropic medication , the dosing of medication must have been kept constant for at least 6 weeks before baseline visit.

Exclusion Criteria:

* Treatment with any antipsychotic medication (neuroleptics) within 8 weeks of baseline visit, or at any time point during the study period.
* Use of tetrabenazine within 12 weeks of baseline visit, or at any time during the study period.
* Treatment with any investigational product within 4 weeks of baseline visit.
* Use of tricyclic antidepressants or class I antiarrhythmics within 6 weeks of baseline visit, or at any time during the study period.
* Use of concomitant medication that may lower the seizure threshold within 6 weeks of baseline visit, or at any time during the study period .
* Use of metoclopramide within 12 weeks of baseline visit, or at any time during the study period.
* Participants currently receiving deep brain stimulation (DBS).
* Participants with a history of surgical procedures aiming to improve the symptoms of Huntington disease, such as neural transplantations, lesions of the central nervous system, infusions of neurotrophic agents or previous attempts of deep brain stimulation.
* Participants previously randomized into this study.
* A prolonged QTc interval at Screening Visit (defined as a QTc interval of > 450 milliseconds [msec] for males or > 470 msec for females), or other clinically significant heart conditions as judged by the investigator.
* Creatinine clearance <40 milliliters (mL)/minute (min) as measured at the screening visit.
* Any clinically significant, abnormal, baseline laboratory result which in the opinion of the Investigator, affects the participant' suitability for the study or puts the participant at risk if he/she enters the study.
* Clinically significant hepatic or renal impairment.
* Participants with a known history of epilepsy or a history of febrile seizure(s) or seizure(s) of unknown cause.
* Severe intercurrent illness, which, in the opinion of the Investigator, may put the participant at risk when participating in the trial or may influence the results of the trial or affect the subjects' ability to take part in the trial.
* Alcohol and/or drug abuse as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM IV-TR) criteria for Substance Abuse - this includes the illicit use of cannabis within the last 12 months prior to Screening Visit
* Participants with suicidal ideation as defined as a positive score on criteria for major depressive episode, item A9 on the DSM -IV-TR criteria for a Major Depressive Episode
* Females who are pregnant or lactating or who intend to become pregnant during the study period.
* Females who are of child bearing potential and not taking adequate contraceptive precautions are excluded from the trial. (Females of childbearing potential taking acceptable contraceptive precautions can be included)
* Known allergy to any ingredients of the trial medication or placebo
* Any previous participation in a clinical study with ACR16.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-10-24 (Actual); Primary Completion 2010-07-26 (Actual); Study Completion 2010-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (28):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, California
  - Colorado Neurological Institute, Littleton, Colorado
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Struthers Parkinson's Center, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - North Shore-LIJ Health System, Manhasset, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Parkinson's Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
- Canada (6):
  - University of Alberta Glenrose Rehab Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - The Centre for Addiction and Mental Health, Markham, Ontario
  - Parkinsons and Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec

REFERENCES:
- [Derived] Darpo B, Geva M, Ferber G, Goldberg YP, Cruz-Herranz A, Mehra M, Kovacs R, Hayden MR. Pridopidine Does Not Significantly Prolong the QTc Interval at the Clinically Relevant Therapeutic Dose. Neurol Ther. 2023 Apr;12(2):597-617. doi: 10.1007/s40120-023-00449-w. Epub 2023 Feb 22. PMID 36811812

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a placebo capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), placebo capsule was taken twice daily (BID) as 2 separate doses.
- ACR16 10 mg BID: Participants received ACR16 10 milligrams (mg) capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 10 mg capsule was taken twice daily (BID) as 2 separate doses (total dose: 20 mg).
- ACR16 22.5 mg BID: Participants received ACR16 22.5 mg capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 22.5 mg capsule was taken twice daily (BID) as 2 separate doses (total dose: 45 mg).
- ACR16 45 mg BID: Participants received ACR16 45 mg capsule once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 45 mg capsule was taken twice daily (BID) as 2 separate doses (total dose: 90 mg).
Period: Overall Study
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Started | 58 | 56 | 55 | 58
Received at Least 1 Dose of Study Drug | 58 | 56 | 55 | 58
Full Analysis Set (All randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization.) | 58 | 55 | 55 | 58
Completed | 55 | 51 | 52 | 55
Not Completed | 3 | 5 | 3 | 3
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 2
Not completed — Investigator decision | 0 | 0 | 1 | 0
Not completed — Did not tolerate study drug | 0 | 0 | 0 | 1
Not completed — Other than specified | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set was defined as all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID | Total
Number analyzed (Participants) | 58 | 55 | 55 | 58 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (10.6) | 54.0 (10.8) | 50.0 (10.5) | 50.3 (9.7) | 51.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 27 | 28 | 120
  Male | 25 | 23 | 28 | 30 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 0 | 2 | 0 | 2 | 4
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 1 | 6
  White | 56 | 52 | 52 | 54 | 214
  More than 1 Race | 0 | 0 | 1 | 1 | 2
Unified Huntington's Disease Rating Scale (UHDRS) Modified Motor Score (mMS) [Mean (Standard Deviation); unit: units on a scale] — The mMS is a subscale of the UHDRS total motor score and comprises 13 responses from the 10 items, 4-10 and 13-15, from the UHDRS motor assessment. The items for mMS included dysarthria, tongue protrusion, finger taps (right and left), pronate/supinate hands (right and left), luria - first-hand-palm sequencing, arms rigidity (right and left), body bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these items were rated on a scale of 0 (normal) to 4 (marked impairment). Total score ranged from 0 to 52, with higher scores indicating more severe motor impairment.
  units on a scale | 17.19 (6.49) | 16.96 (6.18) | 14.18 (5.03) | 16.22 (6.39) | 16.15 (6.13)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Motor Score (mMS) (Sum of Score of Items 4-10 and 13-15 of the UHDRS Motor Assessments) at Week 12
Description: The mMS is a subscale of the UHDRS total motor score and comprises 13 responses from the 10 items, 4-10 and 13-15, from the UHDRS motor assessment. The items for mMS included dysarthria, tongue protrusion, finger taps (right and left), pronate/supinate hands (right and left), luria - first-hand-palm sequencing, arms rigidity (right and left), body bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these items were rated on a scale of 0 (normal) to 4 (marked impairment). Total score ranged from 0 to 52, with higher scores indicating more severe motor impairment. The last observation carried forward (LOCF) method was used to generate an mMS score for each participant for Week 12 assessment.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization. Here, 'Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 53 | 53 | 56
units on a scale | -1.40 (3.72) | -1.30 (3.33) | -2.49 (3.37) | -2.32 (3.72)
Statistical Analysis 1: Comparison: Placebo vs ACR16 45 mg BID; The ANCOVA model included a term for treatment, as well as covariates for baseline mMS, and age at entry to the study; Test type: Superiority; p = 0.078, ANCOVA; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.47 to 0.13]
Statistical Analysis 2: Comparison: Placebo vs ACR16 22.5 mg BID; The ANCOVA model included a term for treatment, as well as covariates for baseline mMS, and age at entry to the study; Test type: Superiority; p = 0.084, ANCOVA — Hypothesis testing was completed only if ACR16 45 mg BID (90 mg) vs. placebo was significant; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-2.53 to 0.16]
Statistical Analysis 3: Comparison: Placebo vs ACR16 10 mg BID; The ANCOVA model included a term for treatment, as well as covariates for baseline mMS, and age at entry to the study; Test type: Superiority; p = 0.982, ANCOVA — Hypothesis testing was completed only if ACR16 22.5 mg BID (45 mg) vs. placebo was significant; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-1.35 to 1.32]

2. Secondary Outcome: Change From Baseline in Total Motor Score (TMS)
Description: The UHDRS Motor Assessment comprises 31 responses from the 15 items, where each response is rated on a 5-point scale from 0 (normal) to 4 (maximally abnormal). The Total Motor Score (TMS) is the sum of all the 31 responses with higher scores indicating more severe motor impairment than lower scores.
Time Frame: Basline, Week 12
Population: The FAS was defined as all randomized participants who received at least 1 dose of study drug and had undergone at least 1 clinical assessment post randomization. Here, 'Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 53 | 53 | 56
Units on a scale | -2.09 (8.31) | -1.92 (6.07) | -3.30 (6.91) | -4.61 (7.21)

3. Secondary Outcome: Number of Participants in Each of the Ratings of the Clinical Global Impression of Change (CGI-C) Scale
Description: The CGI-C was rated by the investigator on a 7-point scale as: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; and 7 = Very much worse.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 55 | 55 | 58
Participants
  Not assessed | 0 | 1 | 1 | 2
  Very much improved | 0 | 1 | 2 | 4
  Much improved | 8 | 3 | 8 | 4
  Minimally improved | 20 | 14 | 17 | 21
  No change | 24 | 31 | 22 | 25
  Minimally worse | 4 | 4 | 5 | 1
  Much worse | 1 | 1 | 0 | 1
  Very much worse | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Stroop Word Reading Test
Description: The Stroop test measures the ability to concentrate and ward off distractions. The test consists of three items: (i) colour naming; (ii) word reading; (iii) interference. The word reading test requires participants to read colour words written in black and each response is scored as the number of correct answers made in 45 seconds. Higher scores indicate less severe disease, and an increase in score represents an improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 55 | 55 | 58
correct responses | 2.5 (13.0) | 3.7 (10.6) | -0.0 (12.7) | 2.8 (10.5)

5. Secondary Outcome: Change From Baseline in Total UHDRS Behavioral Assessment Score
Description: The total behavioral assessment score is the sum of the 11 products (depressed mood, apathy, low self-esteem/guilt, compulsive behavior, anxiety, irritable behavior, perseverative/obsessive thinking, disruptive/aggressive behavior, suicidal thoughts, delusions, and hallucinations) of frequency and severity symptom scores and excluded the 3 yes/no questions relating to confusion, dementia, and depression. Frequency is rated on a scale of 0 (never or almost never) to 4 (very frequently, most of the time). Severity is rated on a scale of 0 (no evidence) to 4 (severe). Total behavior score ranges from 0 (no impairment) to 88 (severe impairment), with higher scores indicating greater behavioral impairments.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 55 | 55 | 58
Units on a scale | -3.56 (8.51) | -3.24 (11.24) | -3.45 (10.10) | -6.19 (10.17)

6. Secondary Outcome: Change From Baseline in Total Hospital Anxiety and Depression Scale (HADS) Score
Description: HADS is a self-administered instrument reliable for detecting states of depression and anxiety. It includes 2 subscales: Hospital Anxiety and Depression Scale - anxiety (HADS-A) assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); Hospital Anxiety and Depression Scale - depression (HADS-D) assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale is comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score ranges from 0 to 21 for each subscale where higher scores indicate greater severity of anxiety and depression symptoms. The total HADS score was a composite score summed of all 14 items for a total range of 0-42. Lower change from baseline scores indicate improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 57 | 55 | 55 | 58
Units on a scale | -1.04 (3.67) | -1.24 (4.57) | -0.95 (4.68) | -2.10 (5.68)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any change from the participant's baseline (pre-treatment) condition, other than improvement, that did not necessarily have causal relationship with the study drug. TEAEs were defined as adverse events that began after ACR16/placebo administration. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ACR16 10 mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Number analyzed (Participants) | 58 | 56 | 55 | 58
Participants | 33 | 30 | 25 | 40

ADVERSE EVENTS:
Time Frame: Baseline up to Week 14
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Adverse events were analyzed for the once a day (first 4 weeks) and twice a day (weeks 5-12) dosing periods and the 2-week follow-up period (up to week 14), as one time period combined per planned analysis for each treatment group.
Groups:
- ACR16 10mg BID: Participants received ACR16 10 milligrams (mg) capsule orally once daily for the first 4 weeks. After 4 weeks (Weeks 5 to 12), ACR16 10 mg capsule was taken twice daily (BID) as 2 separate doses (total dose: 20 mg).
Arm/Group | Placebo | ACR16 10mg BID | ACR16 22.5 mg BID | ACR16 45 mg BID
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/56 | 2/55 | 3/58
Other Adverse Events (participants affected / at risk) | 22/58 | 18/56 | 16/55 | 30/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | ACR16 10mg BID (N=56) | ACR16 22.5 mg BID (N=55) | ACR16 45 mg BID (N=58)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=58) | ACR16 10mg BID (N=56) | ACR16 22.5 mg BID (N=55) | ACR16 45 mg BID (N=58)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 4 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1) | 5 (5)
Fatigue (General disorders) | 5 (6) | 1 (1) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (10) | 9 (10) | 8 (12) | 8 (9)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 3 (3) | 3 (3)
Huntington's chorea (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 30 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 60 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.